CLINICAL TRIAL: NCT03249857
Title: Study of Sensorimotor Compatibility Effects in Bipolar Affective Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1708056; 2017-A00917-46 (Other: ANSM)
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Bipolar Affective Disorder
Keywords: Bipolar affective disorders; Cognition; Emotion; Embodiment; Sensorimotor; Simulation
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Experimental): Patients suffering bipolar affective disorders and who will perform cognitive tasks + IQ + MINI + experimental task
  Interventions: Behavioral: cognitive tasks + IQ + MINI
- control group (Active Comparator): Healthy volunteers (Control group) who will perform cognitive tasks + experimental task
  Interventions: Behavioral: cognitive tasks

INTERVENTIONS:
Behavioral: cognitive tasks + IQ + MINI — Patients will perform different tasks:
  * cognitive tasks : reaction time (Alert TEA, Zimmermann and Fimm, 2005) + Edinburgh laterality questionnaire (Oldfield,1971) + hamilton and young's scale (Tohen et al., 2009) + Montreal Cognitive Assessment (MoCA) (Nasreddine et al., 2005) + experimental task (approach/ avoidance and affordance task).
  * Intelligence Quotient (IQ) test (PM38, Raven, 1960)
  * Mini International Neuropsychiatric Interview (MINI, Van Vliet et al., 2006)
  Arms: patients
Behavioral: cognitive tasks — Healthy volunteers will perform only the cognitive tasks = reaction time alert TEA, Zimmermann and Fimm, 2005 + Edinburgh laterality questionnaire (Oldfield, 1971) + experimental task (approach/ avoidance and affordance task).
  Arms: control group

SUMMARY:
Based in an embodied approach of cognition, several studies have highlighted a direct link between perception of an object or an emotion and the associated motor responses. This study investigated in patients suffering from bipolar affective disorders whether the perception of emotional words involves an automatic sensorimotor simulation of approach and avoidance behaviors, and whether the perception of an object involves an automatic sensorimotor simulation of object prehension (affordance). We hypothesize that, in this pathology, low level (sensorimotor) cognitive processes are preserved whereas high-level (attentional) are altered. 20 patients suffering from bipolar affective disorders and 20 healthy controls will be recruited. The main objective is the emergence of sensorimotor compatibility effects in approach-avoidance task with emotional stimuli (gain between compatible vs incompatible conditions).

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Affiliated or entitled to a social security
* Aged between 18 and 55
* Patients of both sexes suffering from bipolar disorders (DSM V criteria) whatever the subtype
* Stabilized from a point of view clinical and therapeutic
* Euthymic (score <7 at the Hamilton scale, and score <8 at Young's scale)
* Must have given their informed consent before their participation in the study
* Be right-handed (score> 14 on the laterality scale)

For control group:

* Affiliated or entitled to a social security
* Must have given their informed consent before their participation in the study
* Be right-handed (score> 14 on the lateral scale)
* Aged 18 to 55 matched by age (± 5 years), sex, and on the study level of patients (years of schooling after primary school ± 2 years)

Exclusion Criteria:

For patients:

* Thymic acute decompensation
* Hamilton scale > 8, Young's scale > 9
* Montreal Cognitive Assessment (MOCA) <26
* History neurological pathology with cerebral impairment or serious somatic disease
* Disorders related to the use of a psychoactive substance, as defined by the DSM-V (abuse, dependence or withdrawal) within 6 months.
* IQ < 70
* History of head trauma

For control group:

* History of head trauma
* Neurological pathology with cerebral impairment or serious somatic disease
* Psychotropic treatment
* Disorders related to the use of a psychoactive substance, as defined by the DSM-V (abuse, dependence or withdrawal)
* IQ < 70

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
response time for avoidance and affordance task | Months 24
  Comparison of response time for avoidance and affordance task between patients and healthy volunteers.

SECONDARY OUTCOMES:
response time for affordance task | Months 24
  Comparison of response time for affordance task between patients and healthy volunteers.
correlations with age at onset of the disease, the number of thymic decompensations and the existence of psychotic symptoms | Months 24
  These informations were collected of the medical file.
response time and cognitive tests | Months 24
  Correlation between response time and cognitive tests of patients and healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MASSOUBRE, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No